CLINICAL TRIAL: NCT06093464
Title: Beneficial Exposome: Investigating Its Effect on Human Health
Brief Title: Beneficial Exposome Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael Snyder, Professor of Genetics & Genetics Department Chair, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 71135
Record Dates: First submitted 2023-10-04; First posted 2023-10-23 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: All participants will do the intervention but at different times and in different orders.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A- Natural Compound A to Natural Compound B to Natural Compound C (Experimental): * Cycle 1 (4 weeks): use diffused "Natural Compound A" (essential oil) in a diffuser every night when sleeping
  * Cycle 2 (4 weeks): will not use compounds/diffuser (wash-out period)
  * Cycle 3 (4 weeks): use diffused "Natural Compound B" (essential oil) in a diffuser every night when sleeping
  * Cycle 4 (4 weeks): will not use compounds/diffuser (post-intervention observation period)
  * Cycle 3 (4 weeks): use diffused "Natural Compound C" (control) in a diffuser every night when sleeping
  * Cycle 4 (4 weeks): will not use compounds/diffuser (post-intervention observation period)
  There will be 3 natural compounds; the intervention compounds essential oils and are commercially available and there is a control compound (water). They will be used as intended with diffusers.
  Interventions: Other: Natural Compound A (Hinoki essential oil); Other: Natural Compound B (Lemon essential oil); Other: Natural Compound C (Control/Water)
- Group B- Natural Compound B to Natural Compound C to Natural Compound A (Experimental): * Cycle 1 (4 weeks): use diffused "Natural Compound B" (essential oil) in a diffuser every night when sleeping
  * Cycle 2 (4 weeks): will not use compounds/diffuser (wash-out period)
  * Cycle 3 (4 weeks): use diffused "Natural Compound C" (control) in a diffuser every night when sleeping
  * Cycle 4 (4 weeks): will not use compounds/diffuser (post-intervention observation period)
  * Cycle 3 (4 weeks): use diffused "Natural Compound A" (essential oil) in a diffuser every night when sleeping
  * Cycle 4 (4 weeks): will not use compounds/diffuser (post-intervention observation period)
  There will be 3 natural compounds; the intervention compounds essential oils and are commercially available and there is a control compound (water). They will be used as intended with diffusers.
  Interventions: Other: Natural Compound A (Hinoki essential oil); Other: Natural Compound B (Lemon essential oil); Other: Natural Compound C (Control/Water)
- Group C- Natural Compound C to Natural Compound A to Natural Compound B (Experimental): * Cycle 1 (4 weeks): use diffused "Natural Compound C" (control) in a diffuser every night when sleeping
  * Cycle 2 (4 weeks): will not use compounds/diffuser (wash-out period)
  * Cycle 3 (4 weeks): use diffused "Natural Compound A" (essential oil) in a diffuser every night when sleeping
  * Cycle 4 (4 weeks): will not use compounds/diffuser (post-intervention observation period)
  * Cycle 3 (4 weeks): use diffused "Natural Compound B" (essential oil) in a diffuser every night when sleeping
  * Cycle 4 (4 weeks): will not use compounds/diffuser (post-intervention observation period)
  There will be 3 natural compounds; the intervention compounds essential oils and are commercially available and there is a control compound (water). They will be used as intended with diffusers.
  Interventions: Other: Natural Compound A (Hinoki essential oil); Other: Natural Compound B (Lemon essential oil); Other: Natural Compound C (Control/Water)

INTERVENTIONS:
Other: Natural Compound A (Hinoki essential oil) — Participants will use "Natural Compound A" in a diffuser every night for 4 weeks. Diffuser will be placed near participant's bed and will be used during the entire time they are asleep (about 8 hours, every night).
Other: Natural Compound B (Lemon essential oil) — Participants will use "Natural Compound B" in a diffuser every night for 4 weeks. Diffuser will be placed near participant's bed and will be used during the entire time they are asleep (about 8 hours, every night).
Other: Natural Compound C (Control/Water) — Participants will use "Natural Compound C" in a diffuser every night for 4 weeks. Diffuser will be placed near participant's bed and will be used during the entire time they are asleep (about 8 hours, every night).

SUMMARY:
The purpose of this study is to explore the positive, holistic health outcomes resulting from regular exposure to naturally occurring compounds predicted to have health benefits. The researchers hope to learn how the human body is influenced by regular exposure to these compounds.

DETAILED DESCRIPTION:
Considerable research has been conducted on the effects of environmental exposure on human diseases. This is also known as "exposome" research. However, there is limited research on the impact of beneficial exposomes found in the natural environment. The researchers would like to identify and measure the benefits of these naturally occurring compounds on holistic human health.

Through blood specimens, the researchers will observe biomarkers such as cortisol levels and inflammatory markers. Data will be collected from wearable sensors to observe the effects of beneficial exposomes on areas such as cardiovascular health and sleep quality. There will be surveys to understand well-being, stress, and mood. Through such observations, this study aims to understand the positive impacts of intentional exposure to selected compounds found in nature.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Read, speak, and understand English
* Live in the US territory

Exclusion Criteria:

* Mental incapacity and/or cognitive impairment on the part of the patient that would preclude adequate understanding of, or cooperation with, the study protocol
* Is pregnant
* Is breastfeeding
* Has epilepsy
* Has allergies to Cupressaceae family of plants, common plants include redwoods, junipers, cypress, cedar, fir, and sequoia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Resting Heart Rate | Baseline; 26 weeks
  Change in resting heart rate measured by wearable devices
Heart Rate Variability | Baseline; 26 weeks
  Change in resting heart rate measured by wearable devices
Change in sleep quality measured as duration of sleep stages | Baseline; 26 weeks
  Duration of each sleep stage [i.e. light, deep, rapid eye movement (REM), wake stages] overnight. Sleep quality will be measured via a wearable device. Sleep quality will be compared to baseline through the other intervention phases.
Profile of Mood States | Baseline; weeks 2, 6, 10, 14, 18, 22, and 26
  Change in mood states, a 65 item scale that allow for the quick assessment of transient, fluctuating feelings and enduring affect states.

SECONDARY OUTCOMES:
Metabolome | Baseline; weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, and 26
  Change in personal metabolic states as measured in microsampling by targeted and untargeted metabolomics-- liquid chromatography mass spectrometry (LC-MS)-- compared to baseline through the other intervention phases. Dry blood samples will be collected by microsampling bi-weekly at a consistent time in the morning. Based on those samples, metabolomics (e.g., short-chain fatty acids, amino acids and other polar and nonpolar metabolites) will be extracted and quantified by LC-MS.
Proteome | Baseline; weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, and 26
  Comparison of protein changes measured in biospecimens obtained through microsampling against baseline values across various intervention phases. Dry blood samples will be collected by microsampling bi-weekly at a consistent time in the morning. Based on those samples, proteomics will be quantified by proximity extension assay for the cardiometabolic panel. 96 proteins will be measured in the unit of normalized protein expression.
Transcriptome | Baseline; weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, and 26
  Change in messenger ribonucleic acid (mRNA)-based expression measured in biospecimens compared to baseline through the other intervention phases.
Well-being | Baseline; weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, and 26
  Change in well-being measured by Five Well-Being index, a 5-item scale providing a 0 - 25 point composite score, with higher scores indicating greater well-being.
Perceived Stress | Baseline; weeks 2, 6, 10, 14, 18, 22, and 26
  Change in perceived stress measured by Perceived Stress Scale-10, a 10-item scale providing a 0-40 point composite score, with higher scores indicating greater perceived stress.
Generalized Anxiety | Baseline; weeks 2, 6, 10, 14, 18, 22, and 26
  Change in anxiety presence and/or severity measured by Generalized Anxiety Disorder-2, a 2-item scale providing a 0-6 point composite score, with higher scores indicating greater anxiety.
Depression | Baseline; weeks 2, 6, 10, 14, 18, 22, and 26
  Change in depression presence and/or severity measured by Patient Health Questionnaire-2, a 2-item scale providing a 0-6 point composite score, with higher scores indicating greater severity
Inflammation Profile | Baseline; weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, and 26
  Comparison of inflammatory marker changes measured in biospecimens obtained through microsampling against baseline values across various intervention phases. Dry blood samples will be collected by microsampling bi-weekly at a consistent time in the morning. Based on those samples, inflammatory markers will be quantified by targeted 96 Inflammation panel.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Snyder, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.